CLINICAL TRIAL: NCT06738017
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Oral Dose Study Evaluating the Safety and Pharmacokinetics of BMN 349 in Homozygous for the Z Mutation of Alpha 1 Antitrypsin Gene (PiZZ) and Heterozygous for the Z Mutation (PiMZ/MASH)
Brief Title: Study of BMN 349 Single Dose in PiZZ and PiMZ/MASH Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 349-102
Record Dates: First submitted 2024-11-27; First posted 2024-12-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: 349; 349-102; AATD; MASH; PiZZ; PiMZ
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (PiZZ) (Other): 5:1 (349:Placebo)
  Interventions: Drug: BMN 349; Drug: Placebo
- Group B (PiMZ) (Other): 5:1 (349:Placebo)
  Interventions: Drug: BMN 349; Drug: Placebo

INTERVENTIONS:
Drug: BMN 349 — 250mg oral tablet
Drug: Placebo — 250mg oral tablet

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of a single oral dose of BMN 349 in participants with PiZZ or PiMZ/MASH.

Primary outcome measures include incidence of any adverse events (including serious adverse events, dose limit toxicities, and adverse events of special interest), incidence of any laboratory test abnormalities, incidence of lung function test abnormalities and 12-lead ECG parameters.

Participants will receive a single dose of either BMN 349 or placebo and then monitored for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmation of PiZZ or PiMZ genotype
* Females and males, of any race, 18 to 75 years of age
* Nonsmokers, defined as not using tobacco or nicotine-containing products for at least 6 months prior to Screening

Exclusion Criteria:

* International normalized ratio (INR) > 1.2
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 125 U/L
* Current or recent use of AAT augmentation therapy
* Participants with recent (last 3 months) diagnosis of pneumonia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Participant Adverse Events, Serious Adverse Events, Dose Limit Toxicities, Adverse Event of Special Interests, abnormal laboratory tests, abnormal pulmonary function tests, and 12-lead ECG parameters | 78 days
  Number of participant AEs, SAEs, DLTs, AESIs per physician's assessment, abnormal laboratory tests through whole blood samples, abnormal pulmonary function spirometry tests, and 12-lead ECG parameters changes from baseline following a single oral dose of BMN 349

SECONDARY OUTCOMES:
C max | 78 days
  Maximum observed plasma concentration
AUC 0-t | 78 days
  Area under the concentration-time curve from time 0 to the last measurable concentration
AUC 0-inf | 78 days
  Area under the concentration-time curve from time 0 to infinity
CL/F | 78 days
  Apparent total body clearance after oral dosing
T max | 78 days
  Time to reach maximum concentration
t 1/2 | 78 days
  Terminal half-life in plasma
Vz/F | 78 days
  Apparent volume of distribution during terminal phase
Assess functional activity of circulating Alpha1 AntiTrypsin in participants | 78 days
  Changes in participant circulating AAT through whole blood samples following a single dose of BMN 349

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (8):
- United States (4):
  - University of California, San Diego, San Diego, California
  - Saint Louis University, St Louis, Missouri
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - The Medical University of South Carolina, Charleston, South Carolina
- United Kingdom (4):
  - NHS Lothian, Edinburgh, UK
  - Royal Free London NHS Foundation Trust, London, UK
  - Nottingham University Hospitals, Nottingham, UK
  - University Hospital Southampton NHS Foundation Trust, Southampton, UK

IPD SHARING:
Plan to Share IPD: No